CLINICAL TRIAL: NCT02028676
Title: A Randomised Trial of Monitoring Practice and Induction Maintenance Drug Regimens in the Management of Antiretroviral Therapy in Children With HIV Infection in Africa
Brief Title: Efficacy Study of Different Laboratory Management Strategies and Drug Regimens in HIV-infected Children in Africa
Acronym: ARROW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: Department for International Development, United Kingdom (Other Government); ViiV Healthcare (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Diana M Gibb, Professor of Epidemiology, Medical Research Council
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: G0300400; 24791884 (Registry Identifier: ISRCTN); G0300400 (Other Grant/Funding Number: UK Medical Research Council)
Record Dates: First submitted 2013-12-31; First posted 2014-01-07 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Africa; children; antiretroviral therapy; laboratory monitoring; toxicity; CD4; induction maintenance; cotrimoxazole; prophylaxis; abacavir; lamivudine; once daily
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Laboratories; Nevirapine; efavirenz; Zidovudine; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Clinically Driven Monitoring (CDM) (Experimental)
  Interventions: Other: Clinically Driven Monitoring (CDM)
- Laboratory plus Clinical Monitoring (LCM) (Active Comparator)
  Interventions: Other: Laboratory plus Clinical Monitoring (LCM)
- Arm A: abacavir (ABC)+lamivudine (3TC)+NNRTI (Active Comparator): ABC [abacavir]: syrup or tablet, dosed twice-daily according to weight-bands following WHO 3TC [lamivudine]: syrup or tablet, dosed twice-daily according to weight-bands following WHO non-nucleoside reverse transcriptase inhibitor (NNRTI): either nevirapine or efavirenz based on availability (provided by national ART programmes in Uganda/Zimbabwe). Nevirapine syrup or tablet dosed twice-daily according to weight-bands following WHO. Efavirenz tablets dosed once-daily according to weight-bands following WHO.
  Interventions: Drug: Arm A: ABC+3TC+NNRTI
- Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI maintenance (Experimental): ZDV [abacavir]: syrup or tablet, dosed twice-daily according to weight-bands following WHO ABC [abacavir]: syrup or tablet, dosed twice-daily according to weight-bands following WHO 3TC [lamivudine]: syrup or tablet, dosed twice-daily according to weight-bands following WHO NNRTI: either nevirapine or efavirenz based on availability (provided by national ART programmes in Uganda/Zimbabwe). Nevirapine syrup or tablet dosed twice-daily according to weight-bands following WHO. Efavirenz tablets dosed once-daily according to weight-bands following WHO.
  Interventions: Drug: Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI maintenance
- Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC maintenance (Experimental): ZDV [abacavir]: syrup or tablet, dosed twice-daily according to weight-bands following WHO ABC [abacavir]: syrup or tablet, dosed twice-daily according to weight-bands following WHO 3TC [lamivudine]: syrup or tablet, dosed twice-daily according to weight-bands following WHO NNRTI: either nevirapine or efavirenz based on availability (provided by national ART programmes in Uganda/Zimbabwe). Nevirapine syrup or tablet dosed twice-daily according to weight-bands following WHO. Efavirenz tablets dosed once-daily according to weight-bands following WHO.
  Interventions: Drug: Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC maintenance
- Once-daily ABC+3TC (Experimental): ABC [abacavir]: syrup or tablet, dosed once-daily according to weight-bands following WHO 3TC [lamivudine]: syrup or tablet, dosed once-daily according to weight-bands following WHO
  Interventions: Drug: Once-daily ABC+3TC
- Twice-daily ABC+3TC (Active Comparator): ABC [abacavir]: syrup or tablet, dosed twice-daily according to weight-bands following WHO 3TC [lamivudine]: syrup or tablet, dosed twice-daily according to weight-bands following WHO
  Interventions: Drug: Twice-daily ABC+3TC
- Continued cotrimoxazole prophylaxis (Active Comparator): Once-daily doses 5-<15 kg: 200 mg of trimethoprim + 40 mg sulfamethoxazole 15-<30 kg: 400 mg trimethoprim + 80 mg sulfamethoxazole >=30 kg: 800 mg trimethoprim + 160 mg sulfamethoxazole
  Interventions: Drug: Continued cotrimoxazole prophylaxis
- Stopped cotrimoxazole prophylaxis (Experimental): Children had been taking once-daily cotrimoxazole prophylaxis since at least ART initiation. Children randomised to this experimental arm stopped taking cotrimoxazole prophylaxis.
  Interventions: Other: Stopped cotrimoxazole prophylaxis

INTERVENTIONS:
Other: Clinically Driven Monitoring (CDM) — Participants were examined by a doctor and had routine full blood count with white cell differential, lymphocyte subsets (CD4, CD8), biochemistry tests (bilirubin, urea, creatinine, aspartate aminotransferase, alanine aminotransferase) at screening, randomisation (lymphocytes only), weeks 4, 8, and 12, then every 12 weeks. Screening results were used to assess eligibility. All subsequent results at and after randomisation were only returned if requested for clinical management (authorised by centre project leaders); haemoglobin results at week 8 were automatically returned on the basis of early anaemia in a previous adult trial as were grade 4 laboratory toxicities (protocol safety criteria). Total lymphocytes and CD4 tests were never returned for CDM participants, but for all children other investigations (including tests from the routine panels) could be requested and concomitant drugs prescribed, as clinically indicated at extra patient-initiated or scheduled visits.
  Arms: Clinically Driven Monitoring (CDM)
Other: Laboratory plus Clinical Monitoring (LCM) — Participants were examined by a doctor and had routine full blood count with white cell differential, lymphocyte subsets (CD4, CD8), biochemistry tests (bilirubin, urea, creatinine, aspartate aminotransferase, alanine aminotransferase) at screening, randomisation (lymphocytes only), weeks 4, 8, and 12, then every 12 weeks. All results were returned to physicians for patient management. Other investigations (including tests from the routine panels) could be requested and concomitant drugs prescribed, as clinically indicated at extra patient-initiated or scheduled visits.
  Arms: Laboratory plus Clinical Monitoring (LCM)
Drug: Arm A: ABC+3TC+NNRTI — Children received a standard WHO-recommended regimen of open-label lamivudine, abacavir, plus NNRTI continuously. The NNRTI (nevirapine or efavirenz) was chosen by clinicians according to local availability and age.
  Other Names: ABC: abacavir: Ziagen; 3TC: lamivudine: Epivir; ABC+3TC co-formulated: Kivexa; NVP: nevirapine, Viramune; EFV: efavirenz, Sustiva
  Arms: Arm A: abacavir (ABC)+lamivudine (3TC)+NNRTI
Drug: Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI maintenance — Children initiated ART using an induction-maintenance approach, starting with open-label four-drug lamivudine, abacavir, NNRTI, plus zidovudine for 36 weeks, then open-label lamivudine, abacavir, plus NNRTI subsequently. The NNRTI (nevirapine or efavirenz) was chosen by clinicians according to local availability and age.
  Other Names: ZDV: zidovudine, azidothymidine, Retrovir; ABC: abacavir: Ziagen; 3TC: lamivudine: Epivir; ZDV+3TC co-formulated: Combivir; ABC+3TC co-formulated: Kivexa; ZDV+ABC+3TC co-formulated: Trizivir; NVP: nevirapine, Viramune; EFV: efavirenz, Sustiva
  Arms: Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI maintenance
Drug: Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC maintenance — Children initiated ART using an induction-maintenance approach, starting with open-label four-drug lamivudine, abacavir, NNRTI, plus zidovudine for 36 weeks, then open-label lamivudine, abacavir, plus zidovudine subsequently (triple NRTI maintenance). The NNRTI (nevirapine or efavirenz) was chosen by clinicians according to local availability and age.
  Other Names: ZDV: zidovudine, azidothymidine, Retrovir; ABC: abacavir: Ziagen; 3TC: lamivudine: Epivir; ZDV+3TC co-formulated: Combivir; ABC+3TC co-formulated: Kivexa; ZDV+ABC+3TC co-formulated: Trizivir; NVP: nevirapine, Viramune; EFV: efavirenz, Sustiva
  Arms: Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC maintenance
Drug: Once-daily ABC+3TC
  Other Names: ABC: abacavir: Ziagen; 3TC: lamivudine: Epivir; ABC+3TC co-formulated: Kivexa
  Arms: Once-daily ABC+3TC
Drug: Twice-daily ABC+3TC
  Other Names: ABC: abacavir: Ziagen; 3TC: lamivudine: Epivir; ABC+3TC co-formulated: Kivexa
  Arms: Twice-daily ABC+3TC
Drug: Continued cotrimoxazole prophylaxis
  Other Names: trimethoprim+sulfamethoxazole
  Arms: Continued cotrimoxazole prophylaxis
Other: Stopped cotrimoxazole prophylaxis
  Arms: Stopped cotrimoxazole prophylaxis

SUMMARY:
The two original objectives were to determine in HIV-infected children initiating antiretroviral therapy (ART):

1. Whether clinically driven monitoring (CDM) will have a similar outcome in terms of disease progression or death as routine laboratory and clinical monitoring (LCM) for toxicity (haematology/biochemistry) and efficacy (CD4)?
2. Whether induction with four drugs from two ART classes followed by maintenance with three drugs after 36 weeks be more effective than a continuous non-nucleoside reverse transcriptase inhibitors (NNRTI)-based triple drug regimen in terms of CD4 and clinical outcome?

   Two secondary objectives were to determine
3. Whether changing from twice daily lamivudine+abacavir to once daily lamivudine+abacavir after 48 weeks on ART will have a similar outcome in terms of virological suppression and will result in improvements in adherence to ART?
4. Whether stopping daily cotrimoxazole prophylaxis in children over 3 years of age who have been on ART for at least 96 weeks has a similar outcome in terms of hospitalisation or death as continuing daily cotrimoxazole?

DETAILED DESCRIPTION:
The ARROW (AntiRetroviral Research fOr Watoto) protocol describes an open-label randomised trial primarily evaluating two strategic approaches for management of antiretroviral therapy (ART) in 1200 symptomatic HIV-infected infants and children initiating ART following WHO guidelines in Uganda and Zimbabwe. The first strategy compares clinically driven monitoring (CDM) with laboratory plus clinical monitoring (LCM). In both groups, tests for toxicity (standard haematology and biochemistry panels) and efficacy (lymphocyte subsets including CD4 count) will be done every 12 weeks. In LCM, all results will be returned for patient management. In CDM, physicians may request results from routine haematology/biochemistry panels if needed for clinical management, but results will not be returned routinely, and lymphocyte subsets will never be returned. Extra laboratory tests may be requested outside of the scheduled visits at any time in either group (except for lymphocyte subsets in CDM). The second strategy compares a continuous WHO-recommended first-line ART three-drug two-class regimen, comprising two Nucleoside Reverse Transcriptase Inhibitors (NRTIs) plus one Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI), with induction with four drugs (two classes) for 36 weeks followed by maintenance with three drugs. After at least 36 and 96 weeks on ART respectively, two further randomisations will assess simplification strategies which could improve long-term ART adherence (i) once versus twice daily lamivudine+abacavir NRTI drugs (ii) stopping versus continuing daily cotrimoxazole prophylaxis.

ELIGIBILITY:
For initial randomisation to CDM vs LCM, and to ART induction strategy:

Inclusion Criteria:

1. Children should have an adult carer in the household who is either:

   * participating in the DART trial OR
   * being treated with ART OR
   * HIV positive but not yet needing treatment but with access to a treatment programme when ART is required OR
   * HIV negative. Children of DART participants should have first priority on any available remaining slots to enter ARROW.
2. Parents or guardians, and children where appropriate according to age and knowledge of HIV status, must be willing and able to give informed consent for randomisation to CDM or LCM and to first-line ART strategy.
3. Participants must have a confirmed documented diagnosis of HIV-1 infection:

   1. For children aged under 18 months: two separate peripheral blood specimens from different days, both results being positive with HIV-DNA polymerase chain reaction (PCR).
   2. For children aged 18 months or over: antibody positive serology by ELISA test (confirmed by licensed second ELISA or Western Blot) or WHO approved rapid test (performed in series) both on the same sample. Any child previously tested at another clinic should have a repeat test at an ARROW screening laboratory to confirm their status.
4. Age 3 months to 17 years (13-17 years to be capped at 10%)
5. ART naïve (except for exposure to perinatal ART for the prevention of mother-to-child HIV transmission).
6. Meeting criteria for requiring ART according to WHO stage and CD4 percent or count:

   * WHO paediatric clinical stage IV disease: treat regardless of CD4 percent or count
   * WHO paediatric clinical stage III disease:

     * <12 months: treat all
     * >12 months: treat all children irrespective of the CD4 percent or count; however, in children aged > 12 months with tuberculosis, lymphocytic interstitial pneumonia (LIP), oral hairy leukoplakia (OHP) or thrombocytopenia (low platelet count treat) be guided by CD4 cell assays (see below).
   * WHO paediatric clinical stage II or I disease: treat guided by CD4 percent or count

     * CD4%<25% for infants <12 months;
     * CD4%<20% for children 1-<3 years;
     * CD4% <15% for children 3-<5years;
     * CD4% <15% for children > 5years (consideration should also be taken of the CD4 count. A CD4 count <200 cells/mm3 can be used to guide starting ART and CD4 should generally be <350 cells/mm3.)

Exclusion Criteria:

1. Cannot, or unlikely to attend regularly (e.g. usual residence too far from study centre)
2. Likelihood of poor adherence
3. Presence of acute infection (e.g. malaria, helminthiasis, acute hepatitis, acute pneumonia, septicaemia, meningitis). Children may be admitted after recovery of an acute infection. Children with chronic lung disease, including recurrent respiratory infections, are eligible. Children with tuberculosis (TB) will not be enrolled while on the intensive phase of anti-tuberculosis therapy, but should be re-evaluated after the intensive phase and a decision made then about starting ART (see 4 below)
4. In receipt of medication contraindicated by ART

   * children under three years of age receiving anti-tuberculosis therapy should not be enrolled (as they will have to receive nevirapine).
   * on chemotherapy for malignancy
5. Laboratory abnormalities which are a contra-indication for the child to start ART (haemoglobin <8.5g/dL; neutrophils <0.50x109/L; aspartate transaminase (AST) or alanine transaminase (ALT) >5 x the upper limit of normal (ULN); grade 3 renal dysfunction - creatinine >1.9 x ULN).

   N.B. causes of anaemia, such as concurrent bacterial infection, malaria, helminthiasis and/or malnutrition should be investigated, and treatment for anaemia and its causes commenced prior to re-screening for eligibility.
6. Being pregnant or breast-feeding an infant
7. Perinatal exposure to nevirapine (either through prevention of mother-to-child transmission (pMTCT) or breastfeeding) for children aged 3 - 6 months only

Eligibility criteria for the secondary randomisation to once vs twice daily lamivudine+abacavir Inclusion criteria

1. Participating in ARROW
2. On ART for at least 36 weeks
3. Currently taking lamivudine+abacavir twice daily as part of their ART regimen and expected to stay on these two drugs for at least the next 12 weeks
4. Parents or guardians, and children where appropriate according to age and knowledge of HIV status, must be willing and able to give informed consent for randomisation to once or twice daily lamivudine+abacavir

   Exclusion criteria
5. Likely to switch to second-line therapy in the next 12 weeks

Eligibility criteria for the secondary randomisation to stop or continue cotrimoxazole prophylaxis randomisation Inclusion criteria

1. Participating in ARROW
2. Aged at least 3 years
3. Initiated ART at least 96 weeks previously, and received at least 96 weeks of ART allowing for any interruptions in ART
4. Currently prescribed daily cotrimoxazole as primary prophylaxis
5. Parents or guardians, and children where appropriate according to age and knowledge of HIV status, must be willing and able to give informed consent for randomisation to stop or continue daily cotrimoxazole prophylaxis
6. If living in a malaria endemic area, has an insecticide treated bednet and prepared to use this for the child.

   Exclusion criteria
7. Previous diagnosis of Pneumocystis jiroveci pneumonia (cotrimoxazole is secondary prophylaxis and should not be discontinued)

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1206 (Actual)
Dates: Start 2007-03; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Gibb, MD, Principal Investigator — Medical Research Council; Peter Mugyenyi, PhD, Principal Investigator — Joint Clinical Research Centre, Kampala, Uganda; Kusum Nathoo, PhD, Principal Investigator — University of Zimbabwe, Harare, Zimbabwe; Adeodata Kekitiinwa, MD, Principal Investigator — Baylor College of Medicine Children's Foundation, Mulago, Uganda; Paula Munderi, MBChB, Principal Investigator — MRC /UVRI Uganda Research Unit on AIDS, Entebbe, Uganda; Victor Musiime, PhD, Principal Investigator — Joint Clinical Research Centre, Kampala, Uganda; Mutsa F Bwakura-Dangarembizi, MBChB, Principal Investigator — University of Zimbabwe, Harare, Zimbabwe; Philippa Musoke, PhD, Principal Investigator — Baylor College of Medicine Children's Foundation, Mulago, Uganda; Sabrina Bakeera-Kitaka, MBChB, Principal Investigator — Baylor College of Medicine Children's Foundation, Mulago, Uganda; Patricia Nahirya-Ntege, MBChB, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (4):
- Uganda (3):
  - MRC /UVRI Uganda Research Unit on AIDS, Entebbe
  - Joint Clinical Research Centre, Kampala
  - Baylor College of Medicine Children's Foundation, Mulago
- University of Zimbabwe Medical School, Harare, Zimbabwe

REFERENCES:
- [Result] ARROW Trial team. Routine versus clinically driven laboratory monitoring and first-line antiretroviral therapy strategies in African children with HIV (ARROW): a 5-year open-label randomised factorial trial. Lancet. 2013 Apr 20;381(9875):1391-1403. doi: 10.1016/S0140-6736(12)62198-9. Epub 2013 Mar 7. PMID 23473847
- [Result] Bwakura-Dangarembizi M, Kendall L, Bakeera-Kitaka S, Nahirya-Ntege P, Keishanyu R, Nathoo K, Spyer MJ, Kekitiinwa A, Lutaakome J, Mhute T, Kasirye P, Munderi P, Musiime V, Gibb DM, Walker AS, Prendergast AJ. A randomized trial of prolonged co-trimoxazole in HIV-infected children in Africa. N Engl J Med. 2014 Jan 2;370(1):41-53. doi: 10.1056/NEJMoa1214901. PMID 24382064
- [Derived] Musiime V, Kasirye P, Naidoo-James B, Nahirya-Ntege P, Mhute T, Cook A, Mugarura L, Munjoma M, Thoofer NK, Ndashimye E, Nankya I, Spyer MJ, Thomason MJ, Snowden W, Gibb DM, Walker AS; ARROW Trial Team. Once vs twice-daily abacavir and lamivudine in African children. AIDS. 2016 Jul 17;30(11):1761-70. doi: 10.1097/QAD.0000000000001116. PMID 27064996
- See also: main ARROW trial webpage — http://www.arrowtrial.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruited children (n=1206) were randomly assigned to CDM vs LCM and the three different induction ART strategies at enrolment (3/2007-11/2008). This was a factorial randomisation meaning that the children were effectively randomized into 6 parallel groups. Baseline characteristics are presented below separately for each initial randomization.
Pre-assignment Details: There were two additional nested substudy randomizations after initial trial enrolment (see inclusion/exclusion criteria for eligibility). From 8/2009 to 6/2010, eligible children were randomized to once vs twice daily abacavir+lamivudine. From 9/2009 to 2/2011, eligible children were randomized to stop vs continue cotrimoxazole prophylaxis.
Groups:
- Clinically Driven Monitoring (CDM): Clinically Driven Monitoring (CDM): Participants were examined by a doctor and had routine full blood count with white cell differential, lymphocyte subsets (CD4, CD8), biochemistry tests (bilirubin, urea, creatinine, aspartate aminotransferase, alanine aminotransferase) at screening, randomisation (lymphocytes only), weeks 4, 8, and 12, then every 12 weeks. Screening results were used to assess eligibility. All subsequent results were only returned if requested for clinical management (authorised by centre project leaders); haemoglobin results at week 8 were automatically returned on the basis of early anaemia in a previous adult trial as were grade 4 laboratory toxicities (protocol safety criteria). Total lymphocytes and CD4 tests were never returned for CDM participants, but for all children other investigations (including tests from the routine panels) could be requested and concomitant drugs prescribed, as clinically indicated at extra patient-initiated or scheduled visits.
- Once-daily ABC+3TC: ABC [abacavir]: syrup or tablet, dosed once-daily according to weight-bands following WHO 3TC [lamivudine]: syrup or tablet, dosed once-daily according to weight-bands following WHO
  Once-daily ABC+3TC
- Twice-daily ABC+3TC: ABC [abacavir]: syrup or tablet, dosed twice-daily according to weight-bands following WHO 3TC [lamivudine]: syrup or tablet, dosed twice-daily according to weight-bands following WHO
  Twice-daily ABC+3TC
- Continued Cotrimoxazole Prophylaxis: Once-daily doses 5-<15 kg: 200 mg of trimethoprim + 40 mg sulfamethoxazole 15-<30 kg: 400 mg trimethoprim + 80 mg sulfamethoxazole >=30 kg: 800 mg trimethoprim + 160 mg sulfamethoxazole
  Continued cotrimoxazole prophylaxis
- Stopped Cotrimoxazole Prophylaxis: Children had been taking once-daily cotrimoxazole prophylaxis since at least ART initiation. Children randomised to this experimental arm stopped taking cotrimoxazole prophylaxis.
  Stopped cotrimoxazole prophylaxis
Period: Initial Enrolment: CDM vs LCM
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: Abacavir (ABC)+Lamivudine (3TC)+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance | Once-daily ABC+3TC | Twice-daily ABC+3TC | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Started | 606 (Factorial randomization at enrolment: Number of eligible children randomized to this group in ARROW) | 600 (Factorial randomization at enrolment: Number of eligible children randomized to this group in ARROW) | 0 (Factorial randomization at enrolment: Number of eligible children randomized to this group in ARROW) | 0 (Factorial randomization at enrolment: Number of eligible children randomized to this group in ARROW) | 0 (Factorial randomization at enrolment: Number of eligible children randomized to this group in ARROW) | 0 (Secondary partial factorial randomization: Only a subset of ARROW children were eligible) | 0 (Secondary partial factorial randomization: Only a subset of ARROW children were eligible) | 0 (Secondary partial factorial randomization: Only a subset of ARROW children were eligible) | 0 (Secondary partial factorial randomization: Only a subset of ARROW children were eligible)
Completed | 606 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Initial Enrolment: Induction ART
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: Abacavir (ABC)+Lamivudine (3TC)+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance | Once-daily ABC+3TC | Twice-daily ABC+3TC | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Started | 0 | 0 | 397 | 404 | 405 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 397 | 404 | 405 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Subsequent Once vs Twice Daily ABC+3TC
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: Abacavir (ABC)+Lamivudine (3TC)+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance | Once-daily ABC+3TC | Twice-daily ABC+3TC | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Started | 0 | 0 | 0 | 0 | 0 | 336 | 333 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 336 | 333 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Subsequent Cotrimoxazole Randomization
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: Abacavir (ABC)+Lamivudine (3TC)+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance | Once-daily ABC+3TC | Twice-daily ABC+3TC | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 376 | 382
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 376 | 382
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized were included except those who were randomised in error (main enrollment: 1 child HIV-uninfected, 2 on main phase of tuberculosis treatment; cotrimoxazole secondary randomization: 2 children receiving dapsone prophylaxis not cotrimoxazole).
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: Abacavir (ABC)+Lamivudine (3TC)+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance | Once-daily ABC+3TC | Twice-daily ABC+3TC | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis | Total
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405 | 336 | 333 | 376 | 382 | 3839
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age at trial enrollment (antiretroviral therapy initiation).
  years | 5.9 [2.2 to 9.2] | 6.0 [2.6 to 9.4] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 6.0 [2.4 to 9.3]
Age, Customized [Number; unit: participants] — Age at trial enrollment (antiretroviral therapy initiation).
  participants
    < 3 years | 197 | 173 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
    3 years or older | 409 | 427 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 302 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 298 | 298 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants] — Region of enrollment at trial enrollment (antiretroviral therapy initiation).
  participants
    Uganda | 405 | 401 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparisonDifferent randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
    Zimbabwe | 201 | 199 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Age, continuous: Period 2 (trial enrollment, induction ART) [Median (Inter-Quartile Range); unit: years] — Age at trial enrollment (antiretroviral therapy initiation).
  years | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 6.1 [2.4 to 9.3] | 6.2 [2.5 to 9.4] | 5.7 [2.3 to 9.3] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 6.0 [2.4 to 9.4]
Age, continuous: Period 3 (randomization to once vs twice daily ABC+3TC) [Median (Inter-Quartile Range); unit: years] — Age at the time of the secondary randomization to once versus twice daily abacavir+lamivudine (in those children eligible and randomized).
  years | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 5.9 [3.8 to 8.6] | 5.1 [3.6 to 8.3] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 5.5 [3.7 to 8.5]
Age, continuous: Period 4 (randomization to stop versus continue cotrimoxazole) [Median (Inter-Quartile Range); unit: years] — Age at the time of the secondary randomization to stop versus continue cotrimoxazole prophylaxis (in those children eligible and randomized).
  years | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 7.5 [4.6 to 11.1] | 8.3 [4.5 to 11.0] | 7.9 [4.6 to 11.1]
Age, categorical: Period 2 (trial enrollment, induction ART) [Number; unit: participants]
  <3 years | NA — Different randomized comparison | NA — Different randomized comparison | 121 | 117 | 132 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
  3 years or older | NA — Different randomized comparison | NA — Different randomized comparison | 276 | 287 | 273 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Age, categorical: Period 3 (randomization to once vs twice daily ABC+3TC) [Number; unit: participants]
  <3 years | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 36 | 38 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
  3 years and older | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 300 | 295 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Age, categorical: Period 4 (randomization to stop versus continue cotrimoxazole) [Number; unit: participants]
  <3 years | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  3 years and older | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 376 | 382 | NA — Total not calculated because data are not available (NA) in one or more arms.
Gender, Male/Female: Period 2 (trial enrollment, induction ART) [Number; unit: participants]
  Female | NA — Different randomized comparison | NA — Different randomized comparison | 204 | 197 | 209 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Different randomized comparison | NA — Different randomized comparison | 193 | 207 | 196 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Gender, Male/Female: Period 3 (randomization to once vs twice daily ABC+3TC) [Number; unit: participants]
  Female | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 173 | 172 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 163 | 161 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Gender, Male/Female: Period 4 (randomization to stop versus continue cotrimoxazole) [Number; unit: participants]
  Female | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 195 | 203 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparisonDifferent randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 181 | 179 | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment: Period 2 (trial enrollment, induction ART) [Number; unit: participants]
  Uganda | NA — Different randomized comparison | NA — Different randomized comparison | 266 | 268 | 272 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparisonDifferent randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
  Zimbabwe | NA — Different randomized comparison | NA — Different randomized comparison | 131 | 136 | 133 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment: Period 3 (randomization to once vs twice daily ABC+3TC) [Number; unit: participants]
  Uganda | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 249 | 246 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
  Zimbabwe | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparisonDifferent randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 87 | 87 | NA — Different randomized comparison | NA — Different randomized comparison | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment: Period 4 (randomization to stop versus continue cotrimoxazole) [Number; unit: participants]
  Uganda | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 283 | 286 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Zimbabwe | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | NA — Different randomized comparison | 93 | 96 | NA — Total not calculated because data are not available (NA) in one or more arms.
CD4 T cell percentage [Median (Inter-Quartile Range); unit: percentage of total lymphocytes] — CD4 T cell percentage at trial enrollment (antiretroviral therapy initiation).
  percentage of total lymphocytes | 12.5 [7.5 to 17.3] | 12.0 [7.0 to 17.0] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 12.0 [7.3 to 17.1]
CD4 T cell percentage: Period 2 (trial enrollment, induction ART) [Median (Inter-Quartile Range); unit: percentage of total lymphocytes] — CD4 T cell percentage at trial enrollment (antiretroviral therapy initiation).
  percentage of total lymphocytes | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 11.7 [6.9 to 17.5] | 12.0 [7.1 to 17.0] | 12.5 [8.0 to 17.0] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 12.0 [7.3 to 17.1]
CD4 T cell percentage: Period 3 (randomization to once vs twice daily ABC+3TC) [Median (Inter-Quartile Range); unit: percentage of total lymphocytes] — CD4 T cell percentage at the time of the secondary randomization to once versus twice daily abacavir+lamivudine (in those children eligible and randomized).
  percentage of total lymphocytes | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 33.0 [28.0 to 39.0] | 33.0 [27.0 to 39.0] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 33.0 [28.0 to 39.0]
CD4 T cell percentage: Period 4 (randomization to stop versus continue cotrimoxazole) [Median (Inter-Quartile Range); unit: percentage of total lymphocytes] — CD4 T cell percentage at the time of the secondary randomization to stop versus continue cotrimoxazole prophylaxis (in those children eligible and randomized).
  percentage of total lymphocytes | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 33.0 [26.0 to 39.0] | 32.0 [26.0 to 39.0] | 33.0 [26.0 to 39.0]
Duration of antiretroviral therapy: Period 3 (randomization to once vs twice daily ABC+3TC) [Median (Full Range); unit: years] — Years on antiretroviral therapy at the time of the secondary randomization to once versus twice daily abacavir+lamivudine (in those children eligible and randomized).
  years | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 1.8 [0.9 to 3.0] | 1.8 [0.9 to 3.0] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 1.8 [0.9 to 3.0]
Duration of antiretroviral therapy: Period 4 (randomization to stop versus continue cotrimoxazole) [Median (Full Range); unit: years] — Years on antiretroviral therapy at the time of the secondary randomization to stop versus continue cotrimoxazole prophylaxis (in those children eligible and randomized).
  years | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | 2.1 [1.6 to 3.2] | 2.1 [1.8 to 3.2] | 2.1 [1.6 to 3.2]
Weight-for-age Z-score: Period 1 (trial enrollment, CDM vs LCM) [Median (Inter-Quartile Range); unit: Z-score] — Weight-for-age Z-score at trial enrollment (antiretroviral therapy initiation).
  Z-score | -2.3 [-3.4 to -1.3] | -2.2 [-3.3 to -1.3] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | -2.2 [-3.3 to -1.3]
Weight-for-age Z-score: Period 2 (trial enrollment, induction ART) [Median (Inter-Quartile Range); unit: Z-score] — Weight-for-age Z-score at trial enrollment (antiretroviral therapy initiation).
  Z-score | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | -2.3 [-3.5 to -1.3] | -2.2 [-3.2 to -1.4] | -2.2 [-3.4 to -1.3] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | -2.2 [-3.3 to -1.3]
Weight-for-age Z-score: Period 3 (randomization to once vs twice daily ABC+3TC) [Median (Inter-Quartile Range); unit: Z-score] — Weight-for-age Z-score at the time of the secondary randomization to once versus twice daily abacavir+lamivudine (in those children eligible and randomized).
  Z-score | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparisonDifferent randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | -1.4 [-2.0 to -0.7] | -1.3 [-2.0 to -0.6] | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | -1.4 [-2.0 to -0.7]
Weight-for-age Z-score: Period 4 (randomization to stop versus continue cotrimoxazole) [Median (Inter-Quartile Range); unit: Z-score] — Weight-for-age Z-score at the time of the secondary randomization to stop versus continue cotrimoxazole prophylaxis (in those children eligible and randomized).
  Z-score | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | NA [NA to NA] — Different randomized comparison | -1.3 [-1.9 to -0.6] | -1.3 [-1.9 to -0.7] | -1.3 [-1.9 to -0.6]

OUTCOME MEASURES:

1. Primary Outcome: LCM vs CDM: Disease Progression to a New WHO Stage 4 Event or Death
Description: Number of participants with disease progression to a new WHO stage 4 event or death, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Population: All randomized participants (time-to-event)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM)
Number analyzed (Participants) | 606 | 600
participants | 47 | 39
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Non-Inferiority or Equivalence — Upper 95% confidence interval for the hazard ratio was 1.64, see other analysis for this endpoint for details; p = 0.59, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.73 to 1.73] — Hazard ratio is CDM vs LCM
Statistical Analysis 2: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Assumptions: * control group (LCM) event rate 3% per year * rates are reduced to 2% per year in the best of the induction-maintenance arms leading to an overall rate of progression to new WHO stage 4 or death of 2.5% * recruitment is over 1.5 years and follow-up for a minimum further 3.5 years. * cumulative loss to follow-up is 10% at 5 years. See below for rest of sample size as this box is not big enough; Test type: Non-Inferiority or Equivalence — With assumptions detailed above, >90% power and one-sided alpha=0.05, 1160 children would be required to exclude an increase in progression rate of 1.6% from 2.5% to 4.1% per year in the CDM arm (upper 95% confidence limit of LCM: CDM hazard ratio 1.64); p = 0.43, Comparison of poisson rates; Statistical analysis plan specified that p-value was to be calculated from the log-rank test, so not provided for the risk difference; Risk Difference (RD) = 0.32, 95% CI 2-sided [-0.47 to 1.12] — Difference is CDM minus LCM

2. Primary Outcome: LCM vs CDM: New Grade 3 or 4 Adverse Event (AE), Not Solely Related to HIV
Description: Number of participants with a new Grade 3 or 4 adverse event (AE), not solely related to HIV, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM)
Number analyzed (Participants) | 606 | 600
participants | 283 | 282
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.83, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.83 to 1.16] — Hazard ratio is CDM vs LCM

3. Primary Outcome: Induction ART: Change From Baseline in CD4% 72 Weeks After ART Initiation
Time Frame: Baseline, 72 weeks
Population: All participants alive at 72 weeks with CD4 measured (completeness in those in follow-up was 96.6%).
Measure: Mean (Standard Error); unit: percentage of total lymphocytes
Groups:
- Arm A: ABC+3TC+NNRTI: Other Names:
  ABC: abacavir: Ziagen 3TC: lamivudine: Epivir ABC+3TC co-formulated: Kivexa NVP: nevirapine, Viramune EFV: efavirenz, Sustiva Children received a standard WHO-recommended regimen of open-label lamivudine, abacavir, plus NNRTI continuously. The NNRTI (nevirapine or efavirenz) was chosen by clinicians according to local availability and age.
- Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance: Other Names:
  ZDV: zidovudine, azidothymidine, Retrovir ABC: abacavir: Ziagen 3TC: lamivudine: Epivir ZDV+3TC co-formulated: Combivir ABC+3TC co-formulated: Kivexa ZDV+ABC+3TC co-formulated: Trizivir NVP: nevirapine, Viramune EFV: efavirenz, Sustiva Children initiated ART using an induction-maintenance approach, starting with open-label four-drug lamivudine, abacavir, NNRTI, plus zidovudine for 36 weeks, then open-label lamivudine, abacavir, plus NNRTI subsequently. The NNRTI (nevirapine or efavirenz) was chosen by clinicians according to local availability and age.
- Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance: Other Names:
  ZDV: zidovudine, azidothymidine, Retrovir ABC: abacavir: Ziagen 3TC: lamivudine: Epivir ZDV+3TC co-formulated: Combivir ABC+3TC co-formulated: Kivexa ZDV+ABC+3TC co-formulated: Trizivir NVP: nevirapine, Viramune EFV: efavirenz, Sustiva Children initiated ART using an induction-maintenance approach, starting with open-label four-drug lamivudine, abacavir, NNRTI, plus zidovudine for 36 weeks, then open-label lamivudine, abacavir, plus zidovudine subsequently (triple NRTI maintenance). The NNRTI (nevirapine or efavirenz) was chosen by clinicians according to local availability and age
Arm/Group | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 374 | 388 | 374
percentage of total lymphocytes | 16.4 (0.45) | 17.1 (0.43) | 17.3 (0.41)
Statistical Analysis 1: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Assuming a standard deviation for the change in CD4 percentage from baseline to 72 weeks of 10% (slightly higher than that observed in the PENTA 5 trial) 1200 children would provide at least 80% power to detect a difference in change in CD4% from baseline of more than 2.5% across the 3 groups (F-test with 2-sided alpha=0.05) assuming 20% missing data (loss to follow-up during the first year plus failure to attend the week 72 visit/missing sample); Test type: Superiority or Other; p = 0.33, Regression, Linear; Global test with 2df, adjusted for randomization stratification factors

4. Primary Outcome: Induction ART: Change From Baseline in CD4% to 144 Weeks From ART Initiation
Time Frame: Baseline, 144 weeks
Population: All participants alive in follow-up with CD4% (95% completeness)
Measure: Mean (Standard Error); unit: percentage of total lymphocytes
Arm/Group | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 371 | 387 | 378
percentage of total lymphocytes | 19.8 (0.44) | 19.6 (0.49) | 19.2 (0.46)
Statistical Analysis 1: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.69, Regression, Linear; Global test with 2df, adjusted for randomization stratification factors

5. Primary Outcome: Induction ART: New Grade 3 or 4 Adverse Event (AE), Not Solely Related to HIV
Description: as for outcome 2
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Groups:
- ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance: Other Names:
  ZDV: zidovudine, azidothymidine, Retrovir ABC: abacavir: Ziagen 3TC: lamivudine: Epivir ZDV+3TC co-formulated: Combivir ABC+3TC co-formulated: Kivexa ZDV+ABC+3TC co-formulated: Trizivir NVP: nevirapine, Viramune EFV: efavirenz, Sustiva Children initiated ART using an induction-maintenance approach, starting with open-label four-drug lamivudine, abacavir, NNRTI, plus zidovudine for 36 weeks, then open-label lamivudine, abacavir, plus zidovudine subsequently (triple NRTI maintenance). The NNRTI (nevirapine or efavirenz) was chosen by clinicians according to local availability and age
Arm/Group | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 397 | 404 | 405
participants | 157 | 190 | 218
Statistical Analysis 1: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.0001, Log Rank; Global test with 2df, adjusted for randomization stratification factors
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance; Test type: Superiority or Other; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.07 to 1.63] — HR is Arm B vs A
Statistical Analysis 3: Comparison: Arm A: ABC+3TC+NNRTI vs ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.58, 95% CI 2-sided [1.29 to 1.94]

6. Primary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Suppressed HIV RNA Viral Load 48 Weeks After Randomisation
Description: Number of participants with HIV RNA viral load <80 copies/ml at 48 weeks. Measured retrospectively on stored plasma specimens: due to low stored volumes from some children, samples had to be diluted and therefore a threshold of <80 copies/ml was used to indicate suppression.
Time Frame: 48 weeks
Population: All randomized participants with VL result from stored plasma specimen (available for 661/669, 99%, randomized participants)
Measure: Number; unit: participants
Groups:
- Once-daily ABC+3TC; Twice-daily ABC+3TC: Other Names:
  ABC: abacavir: Ziagen 3TC: lamivudine: Epivir ABC+3TC co-formulated: Kivexa
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 330 | 331
participants | 236 | 242
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Non-Inferiority or Equivalence — 631 children would be required to exclude a 12% lower suppression rate in the once daily group with at least 90% power and two-sided alpha=0.05 (lower 95% confidence limit of difference between once and twice daily -12%, the non-inferiority margin). 630 children retains at least 80% (rather than 90%) power to exclude a 10% (rather than 12%) lower suppression rate in the once daily group with one-sided alpha=0.05 (lower 90% confidence limit of difference between once and twice daily -10%); p = 0.65, Chi-squared; Risk Difference (RD) = -1.6, 95% CI 2-sided [-8.4 to 5.2] — Difference in suppression <80 copies/ml in once-daily minus twice-daily

7. Primary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: New Grade 3 or 4 Adverse Event (AE), Not Solely Related to HIV, Judged Definitely/Probably or Uncertain Whether Related to Lamivudine or Abacavir
Description: Number of participants with a new grade 3 or 4 adverse event (AE), not solely related to HIV, judged definitely/probably or uncertain whether related to lamivudine or abacavir, to be analysed using time-to-event methods
Time Frame: Median 2 years (from once vs twice daily randomization to 16 March 2012; maximum 2.6 years)
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
participants | 1 | 0

8. Primary Outcome: Cotrimoxazole: New Hospitalisation or Death
Description: Number of participants with a new hospitalisation or death, to be analysed using time-to-event methods
Time Frame: Median 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Groups:
- Continued Cotrimoxazole Prophylaxis: Other Names:
  trimethoprim+sulfamethoxazole
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 48 | 72
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Assumptions * 5% of children receiving daily cotrimoxazole prophylaxis have a new hospitalisation or death per year * recruitment starts 1 July 2009 with 10% children (those already on ART for >96 weeks) entering immediately, and then the remaining children recruited over the following 15 months as they reach 96 weeks on ART. Follow-up is until March 2012. * cumulative loss to follow-up at March 2012 is 10%. See below for further details as box is not big enough; Test type: Non-Inferiority or Equivalence — With assumptions above, at least 80% power and one-sided alpha=0.05, 947 children would be required in the stop/continue cotrimoxazole prophylaxis comparison to exclude an increase in hospitalisation/death rate of 3% from 5% to 8% per year in the stop cotrimoxazole arm (upper 95% confidence limit of stop:continue hazard ratio 1.6); p = 0.007, Log Rank; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [1.14 to 2.37] — Hazard ratio is stop vs continue
Statistical Analysis 2: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; [analysis description as in outcome 8, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; p = 0.006, Poisson regression for risk difference; Risk Difference (RD) = 4.0, 95% CI 2-sided [0.8 to 7.2] — Risk difference is stop vs continue

9. Primary Outcome: Cotrimoxazole: New Grade 3 or 4 Adverse Event (AE), Not Solely Related to HIV
Description: as for outcome 2
Time Frame: Median 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 55 | 64
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.33, Log Rank; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.83 to 1.72] — Hazard ratio is stop vs continue

10. Secondary Outcome: LCM vs CDM, Induction ART: All-cause Mortality
Description: Number of participants who died from any cause, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
participants | 25 | 29 | 20 | 14 | 20
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.45, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.49 to 1.44] — Hazard ratio is CDM vs LCM
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.43, Log Rank; Global test with 2df, adjusted for randomization stratification factors
Statistical Analysis 3: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance; Test type: Superiority or Other; p = 0.23, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.33 to 1.31] — Hazard ratio is Arm B vs A
Statistical Analysis 4: Comparison: Arm A: ABC+3TC+NNRTI vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.93, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.52 to 1.81] — Hazard ratio is Arm C vs A

11. Secondary Outcome: Induction ART: New WHO Stage 4 Event or Death
Description: Number of participants with a new WHO stage 4 event or death, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 397 | 404 | 405
participants | 30 | 28 | 28
Statistical Analysis 1: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.89, Log Rank; Global test with 2df, adjusted for randomization stratification factors
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance; Test type: Superiority or Other; p = 0.64, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.53 to 1.48] — Hazard ratio is Arm B vs A
Statistical Analysis 3: Comparison: Arm A: ABC+3TC+NNRTI vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.71, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.54 to 1.52] — Hazard ratio is Arm C vs A

12. Secondary Outcome: LCM vs CDM, Induction ART: New WHO Stage 3 or 4 Event or Death
Description: Number of participants with a new WHO stage 3 or 4 event or death, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
participants | 77 | 73 | 73 | 61 | 54
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.98, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.73 to 1.38] — Hazard ratio is CDM vs LCM
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.44, Log Rank; Global test with 2df, adjusted for randomization stratification factors
Statistical Analysis 3: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance; Test type: Superiority or Other; p = 0.30, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.55 to 1.20] — Hazard ratio is Arm B vs A
Statistical Analysis 4: Comparison: Arm A: ABC+3TC+NNRTI vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.24, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.54 to 1.17] — Hazard ratio is Arm C vs A

13. Secondary Outcome: LCM vs CDM, Induction ART: New or Recurrent WHO Stage 3 or 4 Event or Death
Description: Number of participants with a new or recurrent WHO stage 3 or 4 event or death, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
participants | 91 | 79 | 64 | 53 | 53
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.52, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.82 to 1.49] — Hazard ratio is CDM vs LCM
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.34, Log Rank — Global test with 2df, adjusted for randomization stratification factors
Statistical Analysis 3: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance; Test type: Superiority or Other; p = 0.19, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.54 to 1.13] — Hazard ratio is Arm B vs A
Statistical Analysis 4: Comparison: Arm A: ABC+3TC+NNRTI vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.25, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.56 to 1.16] — Hazard ratio is Arm C vs A

14. Secondary Outcome: LCM vs CDM, Induction ART: Weight-for-age Z-score
Description: Age-adjusted change in weight-for-age Z-score at all 12-weekly visits attended over the whole follow-up, no specific timepoint prespecified. Mean and SD are time-averaged area under the change curve calculated using the trapezoidal rule. Z-scores calculated using UK norms which cover the full age range of children (Cole, T. J., J. V. Freeman, and M. A. Preece. 1998. British 1990 growth reference centiles for weight, height, body mass index and head circumference fitted by maximum penalized likelihood. Statistics in Medicine 17(4): 407-29).
Time Frame: Baseline and a median of 4 years (maximum 5 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
age-adjusted z-score | 0.76 (1.05) | 0.78 (1.01) | 0.72 (0.95) | 0.79 (1.00) | 0.80 (1.13)
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.71, Generalized estimating equations; Generalised estimating equations with independent correlation structure and robust standard errors, calculated over all post-randomization visit weeks
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.58, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]

15. Secondary Outcome: LCM vs CDM, Induction ART: Height-for-age Z-score
Description: as for outcome 14
Time Frame: Baseline and a median of 4 years (maximum 5 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
age-adjusted z-score | 0.36 (0.65) | 0.43 (0.66) | 0.40 (0.67) | 0.40 (0.65) | 0.38 (0.64)
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.07, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.90, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]

16. Secondary Outcome: LCM vs CDM, Induction ART: Body Mass Index-for-age Z-score
Description: Age-adjusted change in body mass index-for-age Z-score at all 12-weekly visits attended over the whole follow-up, no specific timepoint prespecified. Mean and SD are time-averaged area under the change curve calculated using the trapezoidal rule. Z-scores calculated using UK norms which cover the full age range of children (Cole, T. J., J. V. Freeman, and M. A. Preece. 1998. British 1990 growth reference centiles for weight, height, body mass index and head circumference fitted by maximum penalized likelihood. Statistics in Medicine 17(4): 407-29).
Time Frame: Baseline and a median of 4 years (maximum 5 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
age-adjusted z-score | 0.65 (1.28) | 0.61 (1.20) | 0.56 (1.11) | 0.64 (1.21) | 0.69 (1.39)
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.64, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.30, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]

17. Secondary Outcome: LCM vs CDM: Change From Baseline in CD4% to Week 72
Time Frame: Baseline, week 72
Population: All participants alive in follow-up with CD4% (97% completeness)
Measure: Mean (Standard Error); unit: percentage of total lymphocytes
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM)
Number analyzed (Participants) | 577 | 563
percentage of total lymphocytes | 17.2 (0.36) | 16.7 (0.35)
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.45, Regression, Linear; Adjusted for randomization stratification factors

18. Secondary Outcome: LCM vs CDM: Change From Baseline in CD4% to Week 144
Time Frame: Baseline, week 144
Population: All participants alive in follow-up with CD4% (95% completeness)
Measure: Mean (Standard Error); unit: percentage of total lymphocytes
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM)
Number analyzed (Participants) | 579 | 557
percentage of total lymphocytes | 19.7 (0.38) | 19.4 (0.38)
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.70, Regression, Linear; Adjusted for randomization stratification factors

19. Secondary Outcome: LCM vs CDM, Induction ART: Change From Baseline in Absolute CD4 to Week 72
Description: Estimated in those >5 years at enrolment, in whom absolute CD4 is meaningful. (In uninfected children, CD4 decreases with age during early childhood.)
Time Frame: Baseline, week 72
Population: All participants alive in follow-up with CD4
Measure: Mean (Standard Error); unit: absolute cells per mm3
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 326 | 325 | 208 | 231 | 212
absolute cells per mm3 | 408 (22.2) | 385 (19.8) | 402 (24.7) | 447 (28.5) | 336 (22.5)
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.59, Regression, Linear; Adjusted for randomization stratification factors
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.01, Regression, Linear; Global test with 2df, adjusted for randomization stratification factors

20. Secondary Outcome: LCM vs CDM, Induction ART: Change From Baseline in Absolute CD4 to Week 144
Description: as for outcome 19
Time Frame: Baseline, week 144
Population: All participants alive in follow-up with CD4
Measure: Mean (Standard Error); unit: absolute cells per mm3
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 326 | 320 | 201 | 231 | 214
absolute cells per mm3 | 418 (20.8) | 420 (22.5) | 446 (25.3) | 450 (28.9) | 360 (24.0)
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.81, Regression, Linear; Adjusted for randomization stratification factors
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.03, Regression, Linear; Global test with 2df, adjusted for randomization stratification factors

21. Secondary Outcome: CDM vs LCM, Induction ART: Suppression of HIV RNA Viral Load 72 Weeks After Baseline
Description: Number of participants with HIV RNA viral load <80 copies/ml 72 weeks after baseline. Threshold for suppression <80 copies/ml as samples had to be diluted due to low volumes.
Time Frame: 72 weeks
Population: Viral loads were assayed retrospectively in a random subset of children
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 98 | 102 | 73 | 85 | 42
participants | 76 | 78 | 56 | 72 | 26
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.86, Chi-squared
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.02, Chi-squared

22. Secondary Outcome: CDM vs LCM, Induction ART: Suppression of HIV RNA Viral Load 144 Weeks After Baseline
Description: Number of participants with HIV RNA viral load <80 copies/ml 144 weeks after baseline. Threshold for suppression <80 copies/ml as samples had to be diluted due to low volumes.
Time Frame: 144 weeks
Population: Viral load was assayed retrospectively at week 144 on a random subset of participants, plus all those aged <5 years at enrolment
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 284 | 266 | 168 | 180 | 203
participants | 192 | 193 | 127 | 135 | 124
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.20, Chi-squared
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.002, Chi-squared

23. Secondary Outcome: LCM vs CDM, Induction ART: Cessation of First-line Regimen for Clinical/Immunological Failure
Description: Number of participants stopping their first-line regimen for clinical/immunological failure, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM)
Number analyzed (Participants) | 606 | 600
participants | 28 | 35
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.22, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.48 to 1.29] — Hazard ratio is CDM vs LCM

24. Secondary Outcome: LCM vs CDM, Induction ART: New Grade 3 or 4 Adverse Event Definitely/Probably or Uncertainly Related to ART
Description: Number of participants with a new grade 3 or 4 adverse event definitely/probably or uncertainly related to ART, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
participants | 30 | 42 | 14 | 30 | 28
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.09, Log Rank; Hazard Ratio (HR) = 0.672, 95% CI 2-sided [0.420 to 1.075] — Hazard ratio is CDM vs LCM
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.04, Log Rank; Global test with 2df, adjusted for randomization stratification factors
Statistical Analysis 3: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance; Test type: Superiority or Other; p = 0.017, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 2.16, 95% CI 2-sided [1.15 to 4.08] — Hazard ratio is Arm B vs A
Statistical Analysis 4: Comparison: Arm A: ABC+3TC+NNRTI vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.034, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 2.00, 95% CI 2-sided [1.05 to 3.80] — Hazard ratio is Arm C vs A

25. Secondary Outcome: LCM vs CDM, Induction ART: New Serious Adverse Events Not Solely Related to HIV
Description: Number of participants with a new serious adverse events not solely related to HIV, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
participants | 147 | 117 | 87 | 82 | 95
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.04, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [1.02 to 1.66] — Hazard ratio is CDM vs LCM
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.53, Log Rank; Global test with 2df, adjusted for randomization stratification factors
Statistical Analysis 3: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance; Test type: Superiority or Other; p = 0.60, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.68 to 1.25] — Hazard ratio is Arm B vs A
Statistical Analysis 4: Comparison: Arm A: ABC+3TC+NNRTI vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.56, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.81 to 1.46] — Hazard ratio is Arm C vs A

26. Secondary Outcome: LCM vs CDM, Induction ART: New ART-modifying Adverse Event
Description: Number of participants with a new ART-modifying adverse event, to be analysed using time-to-event methods
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Number; unit: participants
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
participants | 31 | 32 | 8 | 30 | 25
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.84, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.58 to 1.56] — Hazard ratio is CDM vs LCM
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.002, Log Rank; Global test with 2df, adjusted for randomization stratification factors
Statistical Analysis 3: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance; Test type: Superiority or Other; p = 0.001, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 3.80, 95% CI 2-sided [1.74 to 8.29] — Hazard ratio is Arm B vs A
Statistical Analysis 4: Comparison: Arm A: ABC+3TC+NNRTI vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.006, Regression, Cox; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 3.09, 95% CI 2-sided [1.39 to 6.85] — Hazard ratio is Arm C vs A

27. Secondary Outcome: LCM vs CDM, Induction ART: Adherence to ART as Measured by Self-reported Questionnaire (Missing Any Pills in the Last 4 Weeks)
Description: Binary outcome measure: missed any doses of ART in the last 4 weeks by self-report. Mean calculated across all 12-weekly visits attended over the whole follow-up (no specific timepoint prespecified), giving the percentage of visits attended where the carer/participant reported missing any pills in the last 4 weeks.
Time Frame: Median 4 years (from randomization to 16 March 2012; maximum 5 years)
Measure: Mean (Standard Deviation); unit: % of visits reporting missed pills
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: ABC+3TC+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance
Number analyzed (Participants) | 606 | 600 | 397 | 404 | 405
% of visits reporting missed pills | 8.5 (11.1) | 9.4 (12.4) | 8.3 (10.8) | 9.5 (11.8) | 9.1 (12.7)
Statistical Analysis 1: Comparison: Clinically Driven Monitoring (CDM) vs Laboratory Plus Clinical Monitoring (LCM); Test type: Superiority or Other; p = 0.53, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Arm A: ABC+3TC+NNRTI vs Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance vs Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance; Test type: Superiority or Other; p = 0.46, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]

28. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Suppression of HIV RNA Viral Load 96 Weeks After Randomisation
Description: Number of participants with HIV RNA viral load <80 copies/ml at 96 weeks. Threshold for suppression <80 copies/ml as samples had to be diluted due to low volumes.
Time Frame: 96 weeks
Population: All participants with viral load assayed in stored specimens (98% of those randomized)
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 331 | 326
participants | 230 | 234
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.52, Chi-squared; Risk Difference (RD) = -2.3, 95% CI 2-sided [-9.3 to 4.7]

29. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Change From Baseline in CD4% to Week 48
Time Frame: Randomisation to once vs twice daily, week 48
Population: All participants alive in follow-up with CD4%
Measure: Mean (Standard Deviation); unit: percentage of total lymphocytes
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 331
percentage of total lymphocytes | 0.9 (6.1) | 1.3 (5.4)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.39, Regression, Linear; Adjusted for randomization stratification factors; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.2 to 0.5] — Difference is once-daily minus twice-daily

30. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Change From Baseline in CD4% to Week 72
Time Frame: Baseline, week 72
Population: All participants alive in follow-up with CD4%
Measure: Mean (Standard Deviation); unit: percentage of total lymphocytes
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 332 | 325
percentage of total lymphocytes | 1.9 (6.3) | 1.9 (5.3)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.98, Regression, Linear; Adjusted for randomization stratification factors; Mean Difference (Net) = -0.0, 95% CI 2-sided [-0.9 to 0.9] — Difference is once-daily minus twice-daily

31. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Change From Baseline in CD4% to Week 96
Time Frame: Randomisation to once vs twice daily, week 96
Population: All participants alive in follow-up with CD4%
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 306 | 304
percentage of lymphocytes | 1.6 (7.0) | 2.5 (6.3)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.12, Regression, Linear; Adjusted for randomization stratification factors; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.9 to 0.2] — Difference is once-daily minus twice-daily

32. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Change From Baseline in Absolute CD4 to Week 48
Description: as for outcome 19
Time Frame: Randomisation to once vs twice daily, week 48
Population: All participants aged >5 years at randomization to once versus twice daily alive in follow-up with CD4 measured
Measure: Mean (Standard Deviation); unit: cells per mm3
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 193 | 170
cells per mm3 | 3 (348) | -3 (301)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.82, Regression, Linear; Adjusted for randomization stratification factors; Mean Difference (Net) = 8, 95% CI 2-sided [-60 to 76] — Difference is once-daily minus twice-daily

33. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Change From Baseline in Absolute CD4 to Week 72
Description: All participants aged >5 years at randomization to once versus twice daily alive in follow-up with CD4 measured
Time Frame: Baseline, week 72
Population: All participants aged >5 years at randomization to once versus twice daily alive in follow-up with CD4 measured
Measure: Mean (Standard Deviation); unit: cells per mm3
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 190 | 165
cells per mm3 | -6 (350) | 27 (316)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.36, Regression, Linear; Adjusted for randomization stratification factors; Mean Difference (Net) = -33, 95% CI 2-sided [-104 to 38] — Difference is once-daily minus twice-daily

34. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Change From Baseline in Absolute CD4 to Week 96
Description: All participants aged >5 years at randomization to once versus twice daily alive in follow-up with CD4 measured
Time Frame: Randomisation to once vs twice daily, week 96
Population: All participants aged >5 years at randomization to once versus twice daily alive in follow-up with CD4 measured
Measure: Mean (Standard Deviation); unit: cells per mm3
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 171 | 149
cells per mm3 | -26 (445) | 60 (737)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.20, Regression, Linear; Adjusted for randomization stratification factors; Mean Difference (Net) = -87, 95% CI 2-sided [-220 to 46] — Difference is once-daily minus twice-daily

35. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: All-cause Mortality
Description: Number of participants who died, to be analysed using time-to-event methods
Time Frame: Median 2 years (from randomization to 16 March 2012; maximum 2.6 years)
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
participants | 1 | 4

36. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: New WHO Stage 4 Event or Death
Description: Number of participants with a new WHO stage 4 event or death, to be analysed using time-to-event methods
Time Frame: Median 2 years (from randomization to 16 March 2012; maximum 2.6 years)
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
participants | 3 | 7
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.20, Log Rank; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.11 to 1.64] — Hazard ratio is once-daily vs twice-daily

37. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: New WHO Stage 3 or 4 Event or Death
Description: Number of participants with a new WHO stage 3 or 4 event or death, to be analysed using time-to-event methods
Time Frame: Median 2 years (from randomization to 16 March 2012; maximum 2.6 years)
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
participants | 9 | 12
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.51, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.31 to 1.77] — Hazard ratio is once-daily vs twice-daily

38. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Height-for-age Z-score
Description: Age-adjusted change in height-for-age Z-score over all 12-weekly visits attended over the whole follow-up, no specific timepoint prespecified. Mean and SD are time-averaged area under the change curve calculated using the trapezoidal rule. Z-scores calculated using UK norms which cover the full age range of children (Cole, T. J., J. V. Freeman, and M. A. Preece. 1998. British 1990 growth reference centiles for weight, height, body mass index and head circumference fitted by maximum penalized likelihood. Statistics in Medicine 17(4): 407-29).
Time Frame: Baseline and a median of 2 years (from once vs twice daily randomization to 16 March 2012; maximum 2.6 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
age-adjusted z-score | 0.28 (0.36) | 0.32 (0.45)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.16, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]

39. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Weight-for-age Z-score
Description: as for outcome 14
Time Frame: Baseline and a median of 2 years (from once vs twice daily randomization to 16 March 2012; maximum 2.6 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
age-adjusted z-score | 0.01 (0.35) | -0.00 (0.37)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.54, Generalized estimating equations; [statistical method as in outcome 14, analysis 1]

40. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Body Mass Index-for-age Z-score
Description: as for outcome 16
Time Frame: Baseline and a median of 2 years (from once vs twice daily randomization to 16 March 2012; maximum 2.6 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
age-adjusted z-score | -0.29 (0.49) | -0.35 (0.57)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.08, Generalised estimating equations; [statistical method as in outcome 14, analysis 1]

41. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: New Grade 3 or 4 Adverse Event (AE), Not Solely Related to HIV
Description: as for outcome 2
Time Frame: Median 2 years (from once vs twice daily randomization to 16 March 2012; maximum 2.6 years)
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
participants | 57 | 54
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.82, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.72 to 1.52] — Hazard ratio is once-daily vs twice-daily

42. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: New Serious Adverse Events Not Solely Related to HIV
Description: Number of participants with a new serious adverse event not solely related to HIV, to be analysed using time-to-event methods
Time Frame: Median 2 years (from once vs twice daily randomization to 16 March 2012; maximum 2.6 years)
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
participants | 30 | 37
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.31, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.48 to 1.27] — Hazard ratio is once-daily vs twice-daily

43. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Adherence to ART as Measured by Self-reported Questionnaire (Missing Any Pills in the Last 4 Weeks) at 48 Weeks
Description: Number of participants reporting missing any doses of ART in the last 4 weeks by self-report at 48 weeks.
Time Frame: 48 weeks after randomization to once- versus twice-daily
Population: All participants completing the questionnaire
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 330
participants | 32 | 29
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.74, Chi-squared

44. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Adherence to ART as Measured by Self-reported Questionnaire (Missing Any Pills in the Last 4 Weeks) at 96 Weeks
Description: Number of participants reporting missing any doses of ART in the last 4 weeks by self-report at 96 weeks.
Time Frame: 96 weeks after randomization to once- versus twice-daily
Population: All participants completing the questionnaire
Measure: Number; unit: participants
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 311 | 309
participants | 26 | 25
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.90, Chi-squared

45. Secondary Outcome: Once Versus Twice Daily Abacavir+Lamivudine: Adherence to ART as Measured by Self-reported Questionnaire (Missing Any Pills in the Last 4 Weeks)
Description: as for outcome 27
Time Frame: Mean over median 2 years (from once vs twice daily randomization to 16 March 2012; maximum 2.6 years)
Measure: Mean (Standard Deviation); unit: % of visits reporting missed pills
Arm/Group | Once-daily ABC+3TC | Twice-daily ABC+3TC
Number analyzed (Participants) | 336 | 333
% of visits reporting missed pills | 8 (12) | 8 (12)
Statistical Analysis 1: Comparison: Once-daily ABC+3TC vs Twice-daily ABC+3TC; Test type: Superiority or Other; p = 0.93, Generalized estimating equations; Generalised estimating equation with independent correlation structure and robust standard errors, calculated over all post-randomization visit weeks

46. Secondary Outcome: Cotrimoxazole: New Clinical and Diagnostic Positive Malaria
Description: Number of participants with a new clinical and diagnostic positive malaria, to be analysed using time-to-event methods. Diagnostic positive by either microscopy (thick film) or rapid diagnostic test (RDT)
Time Frame: Median 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 39 | 77
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p < 0.001, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 2.21, 95% CI 2-sided [1.50 to 3.25] — Hazard ratio is stop vs continue

47. Secondary Outcome: Cotrimoxazole: New Severe Pneumonia
Description: Number of participants with a new severe pneumonia, to be analysed using time-to-event methods
Time Frame: Median 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 7 | 10
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.44, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.56 to 3.85] — Hazard ratio is stop vs continue

48. Secondary Outcome: Cotrimoxazole: New WHO Stage 3 or 4 Event or Death
Description: Number of participants with a new WHO stage 3 or 4 event or death, to be analysed using time-to-event methods
Time Frame: Median 2 years (from randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 8 | 19
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.03, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 2.40, 95% CI 2-sided [1.05 to 5.48] — Hazard ratio is stop vs continue

49. Secondary Outcome: Cotrimoxazole: New WHO Stage 3 Severe Recurrent Pneumonia or Diarrhoea
Description: Number of participants with a new WHO stage 3 severe recurrent pneumonia or diarrhoea, to be analysed using time-to-event methods
Time Frame: Median 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 1 | 4
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.18, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 3.98, 95% CI 2-sided [0.44 to 35.7] — Hazard ratio is stop vs continue

50. Secondary Outcome: Cotrimoxazole: New WHO Stage 4 Event or Death
Description: Number of participants with a new WHO stage 4 event or death, to be analysed using time-to-event methods
Time Frame: Median 2 years (from randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 4 | 7
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.34, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.80, 95% CI 2-sided [0.53 to 6.17] — Hazard ratio is stop vs continue

51. Secondary Outcome: Cotrimoxazole: All-cause Mortality
Description: Number of participants who died, to be analysed using time-to-event methods
Time Frame: Median 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 3 | 2
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.68, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.12 to 4.15] — Hazard ratio is stop vs continue

52. Secondary Outcome: Cotrimoxazole: Weight-for-age Z-score
Description: as for outcome 14
Time Frame: Baseline and a median of 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
age-adjusted z-score | -0.01 (0.37) | -0.05 (0.34)
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.07, Generalised estimating equations; [statistical method as in outcome 14, analysis 1]

53. Secondary Outcome: Cotrimoxazole: Height-for-age Z-score
Description: Age-adjusted change in height-for-age Z-score at all 12-weekly visits attended over the whole follow-up, no specific timepoint prespecified. Mean and SD are time-averaged area under the change curve calculated using the trapezoidal rule. Z-scores calculated using UK norms which cover the full age range of children (Cole, T. J., J. V. Freeman, and M. A. Preece. 1998. British 1990 growth reference centiles for weight, height, body mass index and head circumference fitted by maximum penalized likelihood. Statistics in Medicine 17(4): 407-29).
Time Frame: Baseline and a median of 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
age-adjusted z-score | 0.22 (0.33) | 0.19 (0.35)
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.19, Generalised estimating equations; [statistical method as in outcome 14, analysis 1]

54. Secondary Outcome: Cotrimoxazole: Body Mass Index-for-age Z-score
Description: as for outcome 16
Time Frame: Baseline and a median of 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Mean (Standard Deviation); unit: age-adjusted z-score
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
age-adjusted z-score | -0.24 (0.54) | -0.28 (0.45)
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.34, Generalised estimating equations; [statistical method as in outcome 14, analysis 1]

55. Secondary Outcome: Cotrimoxazole: Change From Baseline in CD4% to Week 72
Time Frame: Baseline, week 72
Population: All participants alive in follow-up with CD4%
Measure: Mean (Standard Deviation); unit: percentage of total lymphocytes
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 360 | 360
percentage of total lymphocytes | 1.7 (5.5) | 1.1 (5.7)
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.13, Regression, Linear; Adjusted for randomization stratification factors; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.4 to 0.2] — Difference is stop minus continue

56. Secondary Outcome: Cotrimoxazole: Change From Baseline in Absolute CD4 to Week 72
Description: Estimated in those >5 years at randomization to stop vs continue, in whom absolute CD4 is meaningful. (In uninfected children, CD4 decreases with age during early childhood.)
Time Frame: Baseline, week 72
Population: All participants aged >5 years at randomization to stop versus continue alive in follow-up with CD4 measured
Measure: Mean (Standard Deviation); unit: cells per mm3
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 253 | 254
cells per mm3 | 7 (310) | -2 (303)
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.68, Regression, Linear; Adjusted for randomization stratification factors; Mean Difference (Net) = -11, 95% CI 2-sided [-65 to 42] — Difference is stop minus continue

57. Secondary Outcome: Cotrimoxazole: New Serious Adverse Events Not Solely Related to HIV
Description: as for outcome 42
Time Frame: Median 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Number; unit: participants
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
participants | 32 | 48
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.04, Log Rank; Adjusted for randomization stratification factors; Hazard Ratio (HR) = 1.60, 95% CI 2-sided [1.02 to 2.50] — Hazard ratio is stop vs continue

58. Secondary Outcome: Cotrimoxazole: Adherence to ART as Measured by Self-reported Questionnaire (Missing Any Pills in the Last 4 Weeks)
Description: as for outcome 27
Time Frame: Mean over median 2 years (from cotrimoxazole randomization to 16 March 2012; maximum 2.5 years)
Measure: Mean (Standard Deviation); unit: % of visits reporting missed pills
Arm/Group | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Number analyzed (Participants) | 376 | 382
% of visits reporting missed pills | 9 (13) | 8 (13)
Statistical Analysis 1: Comparison: Continued Cotrimoxazole Prophylaxis vs Stopped Cotrimoxazole Prophylaxis; Test type: Superiority or Other; p = 0.21, Generalised estimating equation — Adjusted for randomization stratification factors; [statistical method as in outcome 45, analysis 1]

ADVERSE EVENTS:
Time Frame: LCM vs CDM and induction-maintenance: median 4 years (maximum 5 years); for randomizations; once vs twice daily: median 2 years (maximum 2.6 years); cotrimoxazole: median 2 years (maximum 2.5 years)
Description: Children were reviewed by a doctor at every scheduled doctor visit, as well as additional visits, and prompts on the doctor follow-up CRF asked about new/worsening/resolved Serious Adverse Events and Grade 3 or 4 Adverse Events.
Arm/Group | Clinically Driven Monitoring (CDM) | Laboratory Plus Clinical Monitoring (LCM) | Arm A: Abacavir (ABC)+Lamivudine (3TC)+NNRTI | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance | Once-daily ABC+3TC | Twice-daily ABC+3TC | Continued Cotrimoxazole Prophylaxis | Stopped Cotrimoxazole Prophylaxis
Serious Adverse Events (participants affected / at risk) | 147/606 | 117/600 | 87/397 | 92/404 | 95/405 | 30/336 | 37/333 | 32/376 | 48/382
Other Adverse Events (participants affected / at risk) | 190/606 | 198/600 | 96/397 | 124/404 | 168/405 | 33/336 | 26/333 | 37/376 | 26/382
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinically Driven Monitoring (CDM) (N=606) | Laboratory Plus Clinical Monitoring (LCM) (N=600) | Arm A: Abacavir (ABC)+Lamivudine (3TC)+NNRTI (N=397) | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance (N=404) | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance (N=405) | Once-daily ABC+3TC (N=336) | Twice-daily ABC+3TC (N=333) | Continued Cotrimoxazole Prophylaxis (N=376) | Stopped Cotrimoxazole Prophylaxis (N=382)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute diarrhoea (Gastrointestinal disorders) | 10 (10) | 6 (6) | 4 (4) | 7 (7) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gasteroenteritis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clinical Anaemia (Blood and lymphatic system disorders) | 17 (18) | 12 (12) | 6 (6) | 10 (11) | 13 (13) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Bronchietasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 6 (6) | 3 (3) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Bone fracture (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Manic psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Trauma (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Hypersensitivity reaction (Skin and subcutaneous tissue disorders) | 22 (22) | 19 (19) | 15 (15) | 15 (15) | 11 (11) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Measles (Infections and infestations) | 7 (7) | 4 (4) | 0 (0) | 5 (5) | 6 (6) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Malaria (Infections and infestations) | 78 (113) | 49 (65) | 48 (69) | 38 (54) | 41 (55) | 19 (27) | 26 (33) | 16 (19) | 34 (47)
Septicaemia/bacteremia (presumptive) (Infections and infestations) | 5 (5) | 5 (6) | 4 (5) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Raised liver enzymes (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis (Hepatobiliary disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm/asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia/arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death, cause unknown (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Death at home with no further information available
Overdose (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal septicaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kwashiorkor (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsions (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinically Driven Monitoring (CDM) (N=606) | Laboratory Plus Clinical Monitoring (LCM) (N=600) | Arm A: Abacavir (ABC)+Lamivudine (3TC)+NNRTI (N=397) | Arm B: ZDV+ABC+3TC+NNRTI->ABC+3TC+NNRTI Maintenance (N=404) | Arm C: ZDV+ABC+3TC+NNRTI->ZDV+ABC+3TC Maintenance (N=405) | Once-daily ABC+3TC (N=336) | Twice-daily ABC+3TC (N=333) | Continued Cotrimoxazole Prophylaxis (N=376) | Stopped Cotrimoxazole Prophylaxis (N=382)
Anaemia with no clinical symptoms (Infections and infestations) | 29 (32) | 37 (41) | 20 (22) | 22 (26) | 24 (25) | 3 (3) | 5 (7) | 5 (5) | 5 (5)
Neutropenia with no clinical symptoms (Investigations) | 151 (211) | 160 (206) | 69 (92) | 105 (138) | 137 (187) | 22 (27) | 15 (16) | 26 (28) | 18 (23)
Thrombocytopenia with no clinical symptoms (Investigations) | 32 (44) | 21 (29) | 19 (24) | 12 (14) | 22 (35) | 9 (15) | 7 (7) | 10 (14) | 6 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No